CLINICAL TRIAL: NCT00271908
Title: Connect to Protect® Partnerships for Youth Prevention Interventions Phase III: Full Evaluation
Brief Title: C2P (With Venues): Connect to Protect® Partnerships For Youth Prevention Interventions
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 040b
Record Dates: First submitted 2005-12-30; First posted 2006-01-04 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-03

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Adolescent; Community; Structural Changes; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort #1: Venue-tracking survey subjects recruited annually for 4 years: N= 320-640 (10-20 members of the population of focus per site, per year). The purpose of this cohort is to identify and track venues at which the population of focus congregates.
  Interventions: Behavioral: Community Mobilization
- Cohort #2: HIV-related risk survey subjects recruited annually for 4 years: N = 1280-2880 (20-30 members of the population of focus per 2-3 congregation venues, per site, per year). These subjects will complete a survey designed to assess HIV-related risk. In the fourth and final year only, HIV Antibody [Ab] assays will also be conducted with survey participants to assess HIV serostatus. The survey and HIVAb assay data will be used to evaluate the intervention within and across sites.
  Interventions: Behavioral: Community Mobilization

INTERVENTIONS:
Behavioral: Community Mobilization — ATN 040b is the evaluation sub-study for ATN 040, Phase III of C2P. Phase III is a community mobilization intervention aimed at reducing HIV rates among youth via community structural change. ATN 040b involves annual anonymous data collection with two cohorts per participating ATN/C2P site. Both cohorts will represent the site's target population, or "population of focus."
  Other Names: No other names

SUMMARY:
During Phase III, Adolescent Trials Network for HIV/AIDS Interventions (ATN)/Connect-to-Protect (C2P) site staff, their official community partners established in Phase I, and newly invited community sector representatives (i.e., individuals from various key parts of the community such as family, spiritual or faith-based institutions, business and government) will form a coalition that will work toward achieving C2P objectives. ATN 040b is the evaluation protocol for ATN 040, Phase III of C2P.

DETAILED DESCRIPTION:
Phase III's objective is to initiate and complete a community mobilization intervention aimed at reducing HIV incidence and prevalence among youth. The intervention will consist of guiding C2P coalitions through a strategic planning process that will result in the development and implementation of a local action plan. The action plan will focus on changing structural elements of the affected communities that are believed to be associated with youth HIV acquisition and transmission. The effectiveness of the intervention will be evaluated by tracking venues where the population of interest congregates and trends in risk factors associated with HIV acquisition and transmission.

ATN 040b evaluates annual anonymous data collection of two cohorts per participating ATN/C2P site. Both cohorts will represent a site's population of focus, but will be recruited in different ways and for different activities.

Cohort #1 will be referred to the site via Official Community Partners and word of mouth. Each year of the study, 10 to 20 individuals will be recruited to complete venue-tracking surveys as described in Section 2.1 (N = 40-80 per site over four years). The results will either confirm that the population of focus can still be reached at previously identified congregation venues or reveal new ones that should be considered for further research activities. Each year, based on data from Cohort #1, ATN/C2P site staff will go to two to three of the confirmed and/or new congregation venues to recruit 20 to 30 participants per venue for Cohort #2. These participants will complete the HIV-related risk survey, with the addition of the HIV-Ab assay in the final year only (N = 160-360 per site over four years). Data will be used to evaluate the intervention within and across ATN/C2P sites.

ELIGIBILITY:
Inclusion Criteria:

* An individual who provides verbal confirmation that his or her age falls within the range of the site's population of focus (which must be within 12 through 24 years, inclusive);
* Verbal confirmation of demographic and sexual orientation/experience profile reflective of the site's population of focus;
* Must report engaging in any voluntary sexual activity (vaginal, anal or oral sex) within the past 12 months, regardless of sexual abuse history; and
* Ability to understand and willingness to provide verbal informed consent/assent in English or Spanish.

Exclusion Criteria:

* Visibly distraught and/or visibly emotionally unstable (e.g., depressive mood; exhibiting manic, suicidal, or violent behavior);*
* Visibly intoxicated or under the influence of psychoactive agents#; or
* Presents as acutely ill.

  * Although it is very unlikely that an individual from the community will overtly show signs of suicidality, youth with any of these exclusion criteria may be approached at a later date if encountered again at the venue and earlier exclusionary conditions are resolved.

    * For sites targeting drug users, this may pose challenges. Potential participants who are visibly under the influence are to be further assessed in terms of their level of alertness, coherency, and abilities to understand and respond to questions. This is to be done keeping staff and participant safety in mind, as well as follow-up procedures such as providing service referrals.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Each site's population of focus was determined during C2P's Phase I (ATN 016a) and is one of the following: young women who have sex with men (YWSM), young men who have sex with men (YMSM), or young users of drugs. For each population, the age range must fall between 12 and 24 years, inclusive.
Sampling Method: Non-Probability Sample
Enrollment: 4472 (Actual)
Dates: Start 2007-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Collect data that will be used to evaluate the overall efficacy of the community mobilization intervention | 4 years
  The aim of ATN 040b is to collect data that will be used to evaluate the overall efficacy of the community mobilization intervention and to assess changes in HIV-related risks over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ellen, MD, Study Chair — Johns Hopkins University
Locations (8):
- United States (7):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Childrens Hospital National Medical Center, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org